CLINICAL TRIAL: NCT02931825
Title: Identification of High Risk People for Colorectal Cancer in Indre-et-Loire (France) and Evaluation of a Specific Surveillance System : a Randomized Trial Assessing the Efficacy of a Letter Encouraging People to Perform Colonoscopy Screening
Brief Title: Identification of High Risk People for Colorectal Cancer and Evaluation of a Specific Surveillance System
Acronym: ISIRECC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: INCa15-SS/ISIRECC; 2015-A01607-42 (Other: ID RCB)
Record Dates: First submitted 2016-10-11; First posted 2016-10-13 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Cancer Colorectal
Keywords: high risk; surveillance; screening; colonoscopy
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reminder letter (Experimental): A letter is sent for remind the importance of compliance with colonoscopy AND to encourage people to to consult their general practitioner or gastroenterologist (if they haven't done their follow-up in time).
  Interventions: Behavioral: Reminder letter
- Control (No Intervention): No intervention (what is done currently)

INTERVENTIONS:
Behavioral: Reminder letter — The letter will consist in several parts:
  * Reminder of : -the need of individual follow-up for high risk people for colorectal cancer AND - the general recommendations (one colonoscopy every 5 years)
  * Recommendation to consult their general practitioner or gastroenterologist if they haven't done their follow up
  * Request information if they've done their follow-up or if we have incorrect information
  * Indication that the letter is sent as part of a surveillance program specific for high risk people for colorectal Cancer
  Arms: Reminder letter

SUMMARY:
Colorectal cancer is one the most frequent cancer in developed countries. In France, it rank third with 43000 new cases in 2015. French Health Authority recommended colonoscopy screening for people with a high risk for colorectal cancer. But this compliance with colonoscopy is low (20-40%), it is therefore necessary to develop new strategies to improve compliance.

The purpose of this project is to to offer and evaluate the feasibility and the effectiveness of a specific surveillance system for high risk people for colorectal cancer

The project will be divided into 2 phases:

Objectives of the first phase:

* Identify high risk people for colorectal cancer in the department of Indre-et-Loire,
* Fill in as completely as possible their colonoscopic history in the past 5 years,
* Estimate the proportion of high risk people for colorectal cancer in the target population for colorectal cancer screening in Indre-et-Loire (Men and women aged from 50 to 74 years).

Objective of the second phase:

Compare the performed colonoscopy rate of high risk people for colorectal cancer without notion of colonoscopy in the past 58 months following or not (control group) the sending of a letter reminding the importance of compliance with colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* residing in Indre et Loire (France)
* with increased risk for colorectal cancer
* who did not perform a colonoscopy in the past 58 months

Exclusion Criteria:

- none

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7101 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2018-05-23 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
Calculate the rate of high risk people for colorectal cancer identified in the target population for colorectal cancer screening in Indre-et-Loire (Men and women aged from 50 to 74 years) | one year
Comparison of the performed colonoscopy rate within 12 months following randomization / send letter in the 2 arms | 12 months after sending the letter (/randomization)

CONTACTS AND LOCATIONS:
Overall Officials: Somany SENGCHANH, Dr, Principal Investigator — Centre de Coordination des Dépistages des Cancers CHRU de Tours; Ken HAGUENOER, Dr, Principal Investigator — Centre de Coordination des Dépistages des Cancers; Julie Boyard, Principal Investigator — Centre de Coordination des Dépistages des Cancers; Thierry Lecomte, Pr, Study Chair — CHRU de Tours, Service Hépato- gastroentérologie
Locations (1):
- UH Tours, Tours, Indre-et-Loire, France

IPD SHARING:
Plan to Share IPD: No